CLINICAL TRIAL: NCT01290029
Title: An Open-label, Single-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Cinacalcet HCl in Pediatric Subjects Aged 28 Days to Less Than 6 Years With Chronic Kidney Disease Receiving Dialysis
Brief Title: Study to Evaluate Cinacalcet in Children With Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20090005
Record Dates: First submitted 2011-01-20; First posted 2011-02-04 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Chronic Kidney Disease; Hyperparathyroidism, Secondary; Secondary Hyperparathyroidism
Keywords: pediatric; CKD; dialysis; paediatric
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary | interventions — Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cinacalcet (Experimental): Participants received a single, oral dose of 0.25 mg/kg cinacalcet.
  Interventions: Drug: Cinacalcet

INTERVENTIONS:
Drug: Cinacalcet — Single, oral dose of 0.25 mg/kg cinacalcet
  Other Names: Sensipar®; Mimpara®

SUMMARY:
The primary objective of the study was to evaluate the safety and tolerability of cinacalcet after a single oral dose in children aged 28 days to less than 6 years with chronic kidney disease receiving dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent, or legally acceptable guardian, must sign an Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved Informed Consent Form.
* Subjects 28 days to < 6 years of age with chronic kidney disease (CKD) and secondary hyperparathyroidism (sHPT) as diagnosed by principal investigators, undergoing hemodialysis or peritoneal dialysis at the time of screening (subjects 6 months or older should have been receiving dialysis for ≥ 1 months) and who have not received any cinacalcet HCl therapy for at least 2 weeks prior to dosing on Day 1
* Free of any disease or condition (other than those diseases or conditions related to their renal disease that, in the opinion of the investigator, would impact the subject's safety or the integrity of the study data).
* Must weigh ≥ 6 kg at screening and at Day-1.
* Must be at least 30 weeks of gestational age.
* Physical examination must be acceptable to the investigator at screening and at Day -1.
* Hemoglobin ≥ 8 g/dL at screening and at Day -1.
* Serum calcium within age-appropriate normal ranges per the National Kidney Foundation Kidney Disease Outcomes Quality Initiative (NKF KDOQI) guidelines at screening and at Day -1
* Normal or clinically acceptable electrocardiogram (ECG) (12-lead reporting RR, PR, QRS, and QTc intervals) at screening and at Day -1.
* Clinical laboratory tests that are acceptable to the investigator at screening and at Day -1.

Exclusion Criteria

* Current or historic malignancy.
* Cardiac ventricular arrhythmias within 28 days prior to screening.
* A gastrointestinal disorder or surgery that could affect the absorption of drugs (eg, pyloric stenosis or any gut-shortening surgical procedure prior to screening).
* A new onset of seizure or worsening of a pre-existing seizure disorder within 2 months prior to IP administration.
* Major surgery (defined as any surgical procedure that involves general anesthesia or respiratory assistance) within 28 days prior to screening.
* Hepatic impairment indicated by elevated levels of hepatic transaminase or bilirubin (aspartate aminotransferase (AST) ≥ 1.5 x upper limit of normal (ULN) OR alanine aminotransferase (ALT) ≥ 1.5 x ULN OR total bilirubin ≥ 1 x ULN per institutional laboratory range) at screening or Day-1.
* History of prolongation of the QT interval (eg, congenital long QT interval, second or third degree heart block or other conditions which prolong the QT interval)
* Corrected QT Interval (QTc) > 500 ms during screening, using Bazett's formula
* QTc ≥ 450 and ≤ 500 ms during screening, using Bazett's formula, unless written permission to enroll is provided by the investigator after consultation with a pediatric cardiologist
* Known hypersensitivity to cinacalcet HCl or any of the excipients in cinacalcet HCl.
* Use of grapefruit juice, herbal medications or potent CYP 3A4 inhibitors (eg, erythromycin, clarithromycin, ketokonazole, itraconazole) within the 14 days prior to enrollment and during the study.
* Concurrent or within 28 days prior to enrollment use of medications that are predominantly metabolized by the enzyme CYP2D6 and have a narrow therapeutic index (eg, flecainide, vinblastine, thioridazine, tricyclic antidepressants such as desipramine and imipramine, and beta-blockers such as metoprolol or carvedilol).
* Concurrent or within 28 days prior to enrollment use of medications that prolong QT interval (eg, sotalol, amiodarone, erythromycin, or clarithromycin).
* Currently receiving treatment in another investigational device or drug study, or less than 90 days since ending treatment on another investigational device or drug study(s).
* Other investigational procedures while participating in this study are excluded.

Ages: 28 Days to 2190 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2011-01-25 (Actual); Primary Completion 2015-09-23 (Actual); Study Completion 2015-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (10):
- United States (4):
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Louisville, Kentucky
  - Research Site, Kansas City, Missouri
- Research Site, Heidelberg, Germany
- United Kingdom (5):
  - Research Site, Bristol
  - Research Site, Glasgow
  - Research Site, Leeds
  - Research Site, Manchester
  - Research Site, Nottingham

REFERENCES:
- [Background] Chen P, Sohn W, Narayanan A, Gisleskog PO, Melhem M. Bridging adults and paediatrics with secondary hyperparathyroidism receiving haemodialysis: a pharmacokinetic-pharmacodynamic analysis of cinacalcet. Br J Clin Pharmacol. 2019 Jun;85(6):1312-1325. doi: 10.1111/bcp.13900. Epub 2019 Apr 25. PMID 30756425
- [Background] Sohn WY, Portale AA, Salusky IB, Zhang H, Yan LL, Ertik B, Shahinfar S, Lee E, Dehmel B, Warady BA. An open-label, single-dose study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of cinacalcet in pediatric subjects aged 28 days to < 6 years with chronic kidney disease receiving dialysis. Pediatr Nephrol. 2019 Jan;34(1):145-154. doi: 10.1007/s00467-018-4054-8. Epub 2018 Aug 23. PMID 30141180
- [Background] Warady BA, Ng E, Bloss L, Mo M, Schaefer F, Bacchetta J. Cinacalcet studies in pediatric subjects with secondary hyperparathyroidism receiving dialysis. Pediatr Nephrol. 2020 Sep;35(9):1679-1697. doi: 10.1007/s00467-020-04516-4. Epub 2020 May 4. PMID 32367309
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 study centers in Belgium (1 site), Germany (1 site), the United Kingdom (2 sites), and the United States (3 sites). The first participant was enrolled 25 January 2011 and the last participant on 25 August 2015.
Pre-assignment Details: Due to blood volume collection limitations in children, participants were randomized in a 1:1 ratio to one of the following 2 pharmacodynamic (PD) sampling sequences: 2, 8, and 48 hours postdose; or 2, 12, and 48 hours postdose.
Groups:
- Cinacalcet 0.25 mg/kg: Participants were to receive a single oral dose of 0.25 mg/kg cinacalcet on day 1.
Period: Overall Study
Arm/Group | Cinacalcet 0.25 mg/kg
Started | 14
Received Study Treatment | 12
Completed | 12
Not Completed | 2
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Cinacalcet 0.25 mg/kg
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: months] | 39.5 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Black (or African American) | 0
  Native Hawaiian or Other Pacific Islander | 0
  White | 9
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: A serious adverse event is defined as an adverse event that meets at least 1 of the following serious criteria: • fatal • life threatening • requires in patient hospitalization or prolongation of existing hospitalization • results in persistent or significant disability/incapacity • congenital anomaly/birth defect • other medically important serious event. Treatment-related adverse events are those the investigator assessed as being possibly related to any study mandated activity (eg, administration of investigational product, protocol-required therapies, device(s) and/or procedure). Events of interest included acute pancreatitis, convulsions, drug related hepatic disorders, fractures, hypersensitivity, hypocalcemia, ischaemic heart disease, ventricular tachyarrhythmias, cardiac failure, and hypotension.
Time Frame: Day 1 to day 30
Population: All participants who received at least 1 dose of cinacalcet.
Measure: Number; unit: participants
Groups:
- Cinacalcet 0.25 mg/kg: Participants received a single oral dose of 0.25 mg/kg cinacalcet on day 1.
Arm/Group | Cinacalcet 0.25 mg/kg
Number analyzed (Participants) | 12
participants
  Any adverse event (AE) | 3
  Serious adverse events | 0
  AE leading to discontinuation of study drug | 0
  Fatal adverse events | 0
  Treatment-related adverse events | 1
  Adverse events of interest | 1

2. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast) for Cinacalcet
Time Frame: Baseline (predose) and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: Pharmacokinetics analysis set
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cinacalcet 0.25 mg/kg
Number analyzed (Participants) | 12
hr*ng/mL | 11.8 (8.74)

3. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUCinf) for Cinacalcet
Time Frame: Baseline (predose) and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: Pharmacokinetics analysis set; The AUCinf value for one participant was excluded based on the goodness-of-fit (R²) value exclusion criteria.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cinacalcet 0.25 mg/kg
Number analyzed (Participants) | 11
hr*ng/mL | 11.3 (7.86)

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Cinacalcet
Time Frame: Baseline (predose) and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: Pharmacokinetics analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cinacalcet 0.25 mg/kg
Number analyzed (Participants) | 12
ng/mL | 2.83 (1.98)

5. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration of Cinacalcet (Tmax)
Time Frame: Baseline (predose) and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: Pharmacokinetics analysis set
Measure: Median (Full Range); unit: hours
Arm/Group | Cinacalcet 0.25 mg/kg
Number analyzed (Participants) | 12
hours | 1.0 (0.820) [0.50 to 4.0]

6. Secondary Outcome: Terminal Half-life of Cinacalcet
Description: The terminal half-life (T1/2) of cinacalcet associated with the slope of the terminal phase.
Time Frame: Baseline (predose) and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: Pharmacokinetics analysis set; The T1/2 value for one participant was excluded based on the goodness-of-fit (R²) value exclusion criteria.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cinacalcet 0.25 mg/kg
Number analyzed (Participants) | 11
hours | 3.70 (2.57)

7. Secondary Outcome: Percent Change From Baseline in Intact Parathyroid Hormone
Time Frame: Baseline (predose) and at 2, 8, 12 and 48 hours post-dose.
Population: Due to the randomization to 1 of 2 sampling sequences not all participants had PD samples taken at every time point. "n" indicates participants with non-missing data at the time point of interest.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Cinacalcet 0.25 mg/kg
Number analyzed (Participants) | 12
percent change
  2 hours post-dose (n = 9) | -10.80 [-18.50 to 23.10]
  8 hours post-dose (n = 5) | -29.6 [-42.20 to -12.60]
  12 hours post-dose (n = 5) | 29.40 [27.70 to 31.20]
  48 hours post-dose (n = 9) | -5.40 [-42.30 to 69.00]

8. Secondary Outcome: Percent Change From Baseline in Total Calcium
Time Frame: Baseline (predose) and 2, 8, 12 and 48 hours post-dose.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cinacalcet 0.25 mg/kg
Number analyzed (Participants) | 12
percent change
  2 hours post-dose (n = 11) | -4.33 (6.82)
  8 hours post-dose (n = 5) | -6.38 (5.12)
  12 hours post-dose (n = 6) | -6.63 (5.05)
  48 hours post-dose (n = 8) | -4.54 (5.12)

9. Secondary Outcome: Percent Change From Baseline in Albumin Corrected Calcium
Time Frame: Baseline (predose) and 2, 8, 12 and 48 hours post-dose.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cinacalcet 0.25 mg/kg
Number analyzed (Participants) | 12
percent change
  2 hours post-dose (n = 9) | -4.01 (7.11)
  8 hours post-dose (n = 5) | -7.12 (6.71)
  12 hours post-dose (n = 5) | -4.24 (1.70)
  48 hours post-dose (n = 6) | -4.10 (5.75)

10. Secondary Outcome: Percent Change From Baseline in Ionized Calcium
Time Frame: Baseline (predose) and 2, 8, 12 and 48 hours post-dose.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cinacalcet 0.25 mg/kg
Number analyzed (Participants) | 12
percent change
  2 hours post-dose (n = 9) | -1.77 (3.55)
  8 hours post-dose (n = 4) | -4.20 (3.83)
  12 hours post-dose (n = 4) | -4.15 (10.12)
  48 hours post-dose (n = 6) | -1.45 (4.80)

ADVERSE EVENTS:
Time Frame: 30 Days
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Cinacalcet 0.25 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cinacalcet 0.25 mg/kg (N=12)
Vomiting (Gastrointestinal disorders) | 1
Catheter site haemorrhage (General disorders) | 1
Device expulsion (General disorders) | 1
Body temperature increased (Investigations) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.